CLINICAL TRIAL: NCT01023191
Title: A Prospective Randomized Controlled Trial of Local Anaesthetic Percutaneous Insertion Versus General Anaesthetic Open Surgical Placement of Continuous Peritoneal Dialysis Catheters in a University Teaching Hospital
Brief Title: Open Versus Percutaneous Insertion of CAPD Catheters
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Did not pass set-up phase
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Collaborators: University of Hull (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Access 3
Record Dates: First submitted 2009-12-01; First posted 2009-12-02 (Estimated); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Renal Failure
Keywords: Dialysis; Peritoneal; Catheter; Surgery
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Percutaneous insertion (Active Comparator): To undergo insertion of catheter using percutaneous technique under local anaesthetic
  Interventions: Procedure: Percutaneous Insertion catheter
- Open insertion (Active Comparator): To undergo insertion of catheter using open technique under general anaesthetic
  Interventions: Procedure: Open insertion Catheter

INTERVENTIONS:
Procedure: Percutaneous Insertion catheter — Insertion of CAPD catheter using percutaneous seldinger technique under local anaesthetic +/- sedation as required
  Arms: Percutaneous insertion
Procedure: Open insertion Catheter — Present technique of open insertion under general anaesthetic. Incision to lower abdomen and direct visualisation of catheter tip placement into pelvis.
  Arms: Open insertion

SUMMARY:
Healthy kidneys clean your blood by removing excess fluid, minerals, and wastes. When your kidneys fail, harmful wastes build up in your body and your body may retain excess fluid. When this happens, you need treatment to replace the work of your failed kidneys. This may be with a dialysis machine using haemodialysis or with fluid in the abdomen or peritoneal dialysis.

In peritoneal dialysis, a tube called a catheter is put in the abdomen wall and used to fill your abdomen with a cleansing liquid called dialysis solution. The walls of your abdominal cavity are lined with a membrane called the peritoneum, which allows waste products and extra fluid to pass from your blood into the dialysis solution. These wastes and fluid are removed from the body when the dialysis fluid is drained and replaced with a fresh solution.

The tubes or catheters used to exchange the fluid are currently positioned using a general anaesthetic (with the patient awake) and an operation with a cut under the belly button. Newer techniques using local anaesthetic (with the patient awake and the area numbed) and requiring only a small cut in the skin have been used. No one has ever directly compared the two techniques.

The investigators aim is to perform a direct comparison between the two techniques to look at the complications and time required for surgery and length of hospital stay required. The investigators will also look at the patients satisfaction and pain scores with each technique to help gather evidence as to which is likely to be the best technique to use from now on.

ELIGIBILITY:
Potential participating patients will be identified by referral to the vascular surgery department for insertion of CAPD catheter for peritoneal access.

Specific inclusion criteria necessary for invitation to study participation;

* Patients referred to vascular consultants for CAPD catheter insertion

General inclusion criteria:

* Ability to give informed written consent

Specific exclusion criteria:

* Previous abdominal surgery via midline incision
* Unfit for general anaesthetic
* Aged under 18 at time of referral

General exclusion criteria:

* Inability to give informed written consent
* Inability to attend follow up appointments

Withdrawal criteria:

* Patient request
* Patient non compliance with study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-02; Primary Completion 2018-07 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Catheter survival | Ongoing (recorded at 6 month intervals)
  Time to catheter removal for any reason.recorded as percentage inn situ at 6, 12,18,etc months post procedure.

SECONDARY OUTCOMES:
Peri operative complications (bleeding, bowel injury) | 24 hrs post procedure
  All complications occuring at time of procedure and in 24 hours immediately post procedure.
Mechanical Complication (drainage failure, displacement, fluid leak) | ongoing (reported at 30 days and monthly thereafter)
  All mechanical complications recorded during follow up period. Note of timing of complications will be made in results. Early = within 30 days, late = beyond 30 days
Infective complications (exit site, tunnel, peritonitis) | ongoing (reported at 30 days and monthly thereafter)
  All infective complications recorded during follow up period. Note of timing of complications will be made in results. Early = within 30 days, late = beyond 30 days
Operative time | Average of 2 hours post procedure
  Time to complete procedure from start to finish.
Technical Success of placement | Average of 2 hours post procedure
  Assessment of whether a working and useable catheter is in situ at the end of the procedure.
Length of admission | Average of 48 hours post procedure
  Length of admission post procedure according to strict discharge criteria.
Patient reported pain post procedure | 24 hour intervals to 5 days post procedure
  Analgesia and daily pain scoring diaries will be issued to patients post procedure. These will record patient reported pain at 24 hour intervals to 5 days as well as analgesia taken during the same period.
Quality of life assessment by questionnaire | Within 24 hours prior to procedure, and again at both 5 days and 3 months post procedure
Estimated cost of care episode | 3 months post procedure
  Overall estimated cost of admission, procedure, ongoing care of catheter and management of complications arising from catheter or procedure will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Ian C Chetter, MB ChB, Principal Investigator — University of Hull
Locations (1):
- Hull Royal Infirmary, Hull, East Yorkshire, United Kingdom

REFERENCES:
- [Derived] Briggs VR, Jacques RM, Fotheringham J, Maheswaran R, Campbell M, Wilkie ME. Catheter insertion techniques for improving catheter function and clinical outcomes in peritoneal dialysis patients. Cochrane Database Syst Rev. 2023 Feb 22;2(2):CD012478. doi: 10.1002/14651858.CD012478.pub2. PMID 36810986